CLINICAL TRIAL: NCT04301024
Title: Nitrous Oxyde Misuse Among Teenagers Consulting in an Addictology Center Dedicated to Young Drug Users: an Observational Study Led in Montpellier
Brief Title: Nitrous Oxyde Misuse Among Teenagers Consulting in an Addictology Center Dedicated to Young Drug Users in Montpellier
Acronym: NC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0116
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Nitrous Oxide; Drug Abuse
Keywords: screening; spotting
MeSH Terms: conditions — Substance-Related Disorders; Metrorrhagia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nitrous oxide misusers: nitrous oxide misusers among the teenagers consulting in an addictology center dedicated to young drug users in Montpellier
  Interventions: Other: assessing the nitrous oxide misuse

INTERVENTIONS:
Other: assessing the nitrous oxide misuse — assessing the nitrous oxide misuse among teenagers consulting in an addioctology center dedicated to young drug users in montpellier

SUMMARY:
Nitrous oxide gas is used in several application areas : medical as an anesthetic drug ; in food industry as a foaming and a mixing agent ; industrial to speed combustion. It is also misused for its hilarant, euphoric and hallucinogenic effect. For this purpose the gas is transfered in a balloon to be inhaled.

As its effects are briefs, its consumption is often perseived as safe. However, some risks exist and are majorated by the way of use and for some groups of people.

Since 2016, the French observatory of drug and substances addiction (OFDT) describes an increasing misuse of nitrous oxide amoung teenagers and young adults. In november 2019, a french press release alerts on the recent increasing of neurologic side effects related to the misuse of nitrous oxide.

That's why, it seems to be interesting to improve the screening of nitrous oxide abuse, in particular amoung adolescents and young adults.

In our study, the investigators would like to determine the characteristics (social, medical, any drug abuse) of teenagers and young adults who misuse nitrous oxide. Through a questionnaire, the investigators plan to select teenagers and young adults who consult in an addictology center dedicated to young drug consumers in Montpellier. This questionnaire is anonymous. The data will be collected only after obtaining the patient's agreement.

The final goal is to create a tool to help general practitioners in screening young people at risk of nitrous oxyde misuse.

ELIGIBILITY:
Inclusion criteria:

- teenagers and young adults consulting in an addictology center dedicated to young abusers in Montpellier and who agree with being included in the study

Exclusion criteria:

- to refuse to participate to the study

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: teenagers and young adults consulting in an addictology center dedicated to young drug abusers in Montpellier
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
nitrous oxide misuse | 1 day
  Description of Nitrous oxide misuse based to answers of a self report questionnaire

SECONDARY OUTCOMES:
use of other drugs (cannabis, tobacco, alcohol, cocaine, heroine) | 1 day
  the use of other drugs (cannabis, tobacco, alcohol, cocaine, heroine. Use of other drug rated by screening test ( CAST ; AUDIT ; Fagerström)
Assess of the side effect based to answers | 1 day
  Assess of the side effect based to answers of a self report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marion Ambrosino, medical resident, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC